CLINICAL TRIAL: NCT03095404
Title: Optimum Dosage of Intravenous Lidocaine for Post-Operative Pain Control in Patients Undergoing Bariatric Bowel Surgery
Brief Title: Intravenous Lidocaine for Post-Operative Pain Control in Patients Undergoing Bariatric Bowel Surgery
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No funding available.
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2198
Record Dates: First submitted 2017-02-21; First posted 2017-03-29 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Bariatric Surgery Candidate
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Dose Lidocaine (Experimental): 60 cc syringe with 2 vials of 1% lidocaine (40cc's) low dose solution using adjusted body weight formula
  Interventions: Drug: Low Dose Lidocaine
- High Dose Lidocaine (Experimental): 60 cc syringe with 2 vials of 2% lidocaine (40 cc's) high dose solution using adjusted body weight formula
  Interventions: Drug: High Dose Lidocaine

INTERVENTIONS:
Drug: Low Dose Lidocaine — 60 cc syringe with 2 vials of 1% lidocaine (40cc's) low dose solution using adjusted body weight formula
  Other Names: Lidocaine 1% Injectable Solution
  Arms: Low Dose Lidocaine
Drug: High Dose Lidocaine — 60 cc syringe with 2 vials of 2% lidocaine (40 cc's) high dose solution using adjusted body weight formula
  Other Names: Lidocaine 2% Injectable Solution
  Arms: High Dose Lidocaine

SUMMARY:
Currently, there are no studies that address the optimum dosage of lidocaine for surgical procedures. Lidocaine is a local anesthetic that is injected to induce anesthesia. Improper or inefficient pain treatment can lead to longer hospital stay, and adverse side effects such as nausea and vomiting. Opioids are the primary drug to treat moderate to severe pain, but are also responsible for nausea and other side effects. Lidocaine has shown to have opioid sparing effects; meaning less opioid use is necessary for pain relief. In this study, we will conduct a clinical trial to assess the difference between different lidocaine dosage schedules to determine the optimum dosage that brings maximum pain relief while minimizing adverse side effects and patient stay. A large benefit in using lidocaine is its documented opioid sparing which allows for minimal drug treatment.

DETAILED DESCRIPTION:
Lidocaine was first discovered from systematic investigations at the Institute of Chemistry at Stockholm. In the early 1940s, Nils Lofgren discovered lidocaine as a potent anesthetic, initially labelled LL30. It was first clinically tested in 1994, and stood up to appraisal as a reliable and highly efficient local anesthetic.

One systematic review found that, depending on the duration of the infusion of lidocaine, significantly different pain ratings resulted. Similarly, a review found low to moderate evidence for an effect of intravenous lidocaine on pain at rest as one of the major predefined outcomes. Interestingly, this was true for a large variation between the bolus doses (1 to 3mg/kg) and continuous infusion regimes (1.5 to 5 mg/kg/h). The variation of doses impacted pain; early and intermediate, postoperative ileus, time to first flatus, and time to first bowel movements/sounds. One study based all medications in the protocol on the dosing body weight [ideal body weight (IBW) + 0.4 x (actual body weight-IBW). Besides an important improvement in overall quality of recovery, subjects had an improvement in the physical comfort, pain, and physical independence subcomponents of the quality of recovery score. Additionally, there was an opioid sparing effect observed in patients undergoing laparoscopic bariatric surgery, making it especially critical due to the limited respiratory reserve of the bariatric population.

Another study assigned subjects in the experimental group to an IV infusion of 2mg/kg per hour of lidocaine, maintained 15 to 30 minutes before skin closure. The study found similar positive effects, improving postoperative analgesia, reducing postoperative opioid requirements, and accelerating the return of the first flatus. Specifically, the investigation found results similar to previous investigations with longer infusion times across a variety of surgical procedures.

Based on the above, there is a call for further research evaluating the optimum dosage of lidocaine infusion in bariatric populations undergoing major surgery. Not only are there a wide variety of positive effects of lidocaine that need to be investigated, but there is a need for precision and sensitivity of dose regimes in a bariatric population susceptible to adverse effects. It is therefore of interest to find an optimal dosage schedule in order to provide anesthesiologists with a standard which maximizes opioid sparing effects, whilst minimizing patient pain, hospital stay, as well as nausea and vomiting.

Given the complexity of this proposed randomized-controlled trial, as well as time and financial limitations, a pilot study was deemed necessary to find out the feasibility and safety of comparing different dosing schedules, rate of patient recruitment, funding necessities, and needs of additional personnel.

ELIGIBILITY:
Inclusion Criteria:

* Bariatric patients 18 years or older undergoing major bowel surgery
* Patient capable to complete informed consent

Exclusion Criteria:

* Pediatric population
* Inability to complete informed consent
* Patient refusal
* Chronic aspirin or NSAID intake
* Known allergy to aspirin and/or NSAIDs, or lidocaine
* History of bronchial asthma requiring intubation
* Peptic ulceration
* Coagulopathy
* Renal insufficiency
* Opioid abuse
* Pregnancy
* Conversion from laparoscopic to open surgery.
* Other relative contraindications for lidocaine; unstable CAD, Recent MI, Heart Failure, Heart Block, Electrolyte Disturbances, Liver Disease, Cardiac Dysrhythmias, and Seizure Disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Evaluation of an intravenous lidocaine dosing schedule using 1mg/kg or 2mg/kg adjusted body weight | 5 days
  Feasibility and safety of different dosing schedules

SECONDARY OUTCOMES:
Amount of intraoperative narcotics used post-surgery | 1 day
  Morphine equivalents in mg of narcotic used
Pain scores | 2 days
  Using visual analogue scale
Enhancement of gastrointestinal recovery | 24 hours
  Time to first flatus and/or bowel movement and incidence of paralytic ileus
Post-operative nausea and vomiting | 24 hours
  Using 0-4 nausea and vomiting scale
Patient satisfaction | 1 day
  Using American Pain society outcome questionnaire
Time of rescue analgesia | 24 hours
  Time in minutes for participant to request for extra pain medication
Length of stay in recovery room | 1 day
  Time in hours for recovery room stay
Length of hospital stay | 5 days
  Number of days in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Greg Peachey, MD, Principal Investigator — McMaster University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aubrun F, Mazoit JX, Riou B. Postoperative intravenous morphine titration. Br J Anaesth. 2012 Feb;108(2):193-201. doi: 10.1093/bja/aer458. PMID 22250276
- [Background] Han PY, Duffull SB, Kirkpatrick CM, Green B. Dosing in obesity: a simple solution to a big problem. Clin Pharmacol Ther. 2007 Nov;82(5):505-8. doi: 10.1038/sj.clpt.6100381. PMID 17952107